CLINICAL TRIAL: NCT06124287
Title: MR Enterography Predictors of Disease Relapse After Stopping Biologic Therapy in Crohn's Disease (METEOR).
Brief Title: MRE Predictors of Disease Relapse After Stopping Biologics
Acronym: METEOR
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: British Society of Gastrointestinal and Abdominal Radiology (BSGAR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 162205
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn's Disease patients stopping biologic therapy: Crohn's Disease patients stopping biologic therapy and undergoing MR Enterography 3 months before or 1 month after this decision as part of standard clinical care.
  Interventions: Diagnostic Test: MR Enterography (MRE)

INTERVENTIONS:
Diagnostic Test: MR Enterography (MRE) — MRI scan

SUMMARY:
This study aims to investigate if MR Enterography (MRE) improves the ability to predict which Crohn's disease patients will relapse quickly (disease comes back) after stopping biologic medication. MRE is a safe MRI scan of the bowel, widely used in Crohn's disease patients.

DETAILED DESCRIPTION:
This study aims to investigate if MR Enterography (MRE) improves the ability to predict which Crohn's disease patients will relapse (disease comes back) after stopping biologic medication when clinically well. MRE is a safe MRI scan of the bowel, widely used in Crohn's disease patients.

Using a network of British Society of Gastrointestinal and Abdominal Radiology (BSGAR) affiliated NHS hospitals, up to 200 patients who have stopped biologic treatment and recently underwent MRE as part of usual care will be identified. Detailed analysis will be performed on these MRI scans using scores measuring residual bowel inflammation, and retrospectively collect standard clinical data such as blood, stool and colonoscopy results. Using hospital records (accessed by each local care team before being pseudoanonymised) the study will see what happened to patients after one year, specifically if they relapsed or remained well off the biologics.

Based on a literature review, the most promising predictors of early relapse will be identified, such as blood/stool tests, to build a statistical model that provides the risk of a patient relapsing within one year. MRE scores will be added to this model to see if it improves the ability to predict relapse.

The results of the study could form part of a clinical decision support tool to help risk stratify patients and improved joint management decision making.

ELIGIBILITY:
Inclusion Criteria:

* Luminal small bowel or colonic Crohn's disease in clinical remission
* 16 years or older
* MRE as part of routine care performed within three months prior, or one month after the decision to stop biologic therapy Anti-TNF (Adalimumab, infliximab, Certolizumab) IL-23 or IL-12 antagonists (Ustekinumab) Anti-integrin biologics (Natalizumab, Vedolizumab)
* Biologic therapy stopped due to clinical remission only

Definition of clinical remission: There is no agreed consensus on how clinical remission is defined and practice differs between hospitals and patients. To mirror current clinical practice, no strict definition of clinical remission will therefore be used. Detailed clinical parameters the time of stopping biologic agents will be collected.

Exclusion Criteria:

<16 years of age

Non-biological therapy, unless part of combination therapy with biologic agents

Biological therapy stopped for other reasons e.g. loss of effect, side effects

Resection of diseased segment(s) after MRE but before stopping biologic agent.

No MRE with the time window defined by eligibility criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn's disease patients will be identified after the clinical decision to stop biologics including during outpatient clinics, multidisciplinary meetings, any local patient databases, and imaging investigation requests.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To develop and internally evaluate a multivariable prediction model for early disease relapse in patients stopping biological therapy | 1 year prediction
  To develop and internally evaluate a multivariable prediction model for early (within one year) disease relapse in patients stopping biological therapy, combining pre-existing clinical parameters with MRE parameters and compare to a baseline model incorporating clinical variables alone

SECONDARY OUTCOMES:
Establish which individual MRE finding/combination of findings best predicts disease relapse after stopping biologic therapy, including complete transmural healing. | 1 year

OTHER OUTCOMES:
To investigate the association of biologic treatment duration on relapse at one year. | 1 year
To investigate the association of concurrent medication use after stopping biologics on relapse at one year. | 1 year
To establish the most common criteria for diagnosing disease relapse used by multidisciplinary consensus panels. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maira Hameed, Principal Investigator — University College London Centre for Medical Imaging
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided